CLINICAL TRIAL: NCT02790333
Title: A Randomized Trail Of Different Stapler Cartridge For Pancreatic Stump Texture To Prevent Pancreatic Fistula After Laparoscopic Distal Pancreatectomy
Brief Title: Different Stapler Cartridge For Pancreatic Stump Texture To Prevent Pancreatic Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi-Ping Mou (Other)
Responsible Party: Sponsor-Investigator, Yi-Ping Mou, MD，Director, Zhejiang Provincial People's Hospital
Organization: Zhejiang Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZJPPH-04
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Neoplasms; Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tri-Staple reloads (Experimental): Tri-Staple reloads were used for pancreatic stump texture
  Interventions: Procedure: Tri-Staple reloads
- traditional reloads (Active Comparator): the traditional reloads were used for pancreatic stump texture
  Interventions: Procedure: traditional reloads

INTERVENTIONS:
Procedure: traditional reloads — Blue cartridge with3.0mm height staple was used for pancreatic stump
  Arms: traditional reloads
Procedure: Tri-Staple reloads — Purple cartridge with2.0-2.5-3.0mm varied-height staples was used for pancreatic stump
  Arms: Tri-Staple reloads

SUMMARY:
The purpose of this trial is to establish an objective criterion for assessing pancreatic stump texture, and unify stapler cartridge according to pancreatic stump texture and thickness.

DETAILED DESCRIPTION:
Distal pancreatectomy (DP) is the standard treatment for symptomatic benign, premalignant, and malignant lesions in the pancreatic body and tail.Laparoscopic distal pancreatectomy (LDP) are reported to have lower blood loss, fewer postoperative complications and a shorter length of stay without a substantial increase in the operative time. Pancreatic fistula (PF) is the major source of postoperative morbidity and is associated with numerous further complications, suffering, longer hospital stay, higher costs and sometimes death. Frequencies range from 5% to 64%. Several procedures have been proposed to reduce the rate of PF. stapler closure is considered to be safe and approved particularly in LDP. Numerous predictive factors for PF have been reported in previous studies. Among these risk factors, the most important might be the texture and thickness of the remnant pancreas. However, the judgment of pancreatic texture has been based on the surgeon's observation and there still exists no objective method of assessing pancreatic texture. Furthermore there is no strict guideline on which type of cartridge to use according to pancreatic stump texture and thickness. Therefore, this single blind randomized controlled trial is designed to establish an objective criterion for assessing pancreatic stump texture, and unify stapler cartridge according to pancreatic stump texture and thickness. Patients were stratified intraoperatively by gland texture-hard (fibrotic) or soft (normal) and subsequently randomized according to different stapler cartridge. Pancreatic fibrosis is accessed by histopathology and pancreatic stellate cell.

ELIGIBILITY:
Inclusion Criteria:

1. disease of pancreatic body and tail
2. Age: 18 years or older
3. distant metastases are not diagnosed preoperatively.
4. Patients who can provide written informed consent

Exclusion Criteria:

1. Patients with severe organ disease such as cardiac disease,respiratory illness
2. Patients with pancreaticojejunostomy,pancreatogastrostomy
3. Patients with conversion to laparotomy
4. Patients with pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of pancreatic fistula grade A/ B/C defined by ISGPF classification | Thirty days after operation
  Pancreatic amylase concentration in any post operative drains. Fistula is diagnosed if pancreatic amylase > 3 times the upper normal limit of pancreatic amylase in plasma on post operative day 3 or later
Pancreatic fibrosis accessed by histopathology and pancreatic stellate cell | intraoperative

SECONDARY OUTCOMES:
Morbidity | Thirty days after operation
Mortality | Thirty days after operation
Time to oral intake | Duration of hospital stay
Postoperative hospital stay | Duration of hospital stay
Readmission rate | Thirty days after operation

CONTACTS AND LOCATIONS:
Overall Officials: YiPing Mou, MD, Study Director — Department of Gastrointestinal-Pancreatic Surgery, Zhejiang Provincial Peoples' Hospital
Locations (1):
- Zhejiang Provincial Peoples' Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided